CLINICAL TRIAL: NCT06644833
Title: Effectiveness of Transcranial Magnetic Stimulation (TMS) Versus Treatment as Usual for First-Episode Depression in Adult Patients. An Open-Label Randomised Controlled Trial
Brief Title: Effective of Transcranial Magnetic Stimulation (TMS) vs Treatment as Usual for First-Episode Depression in Adults
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Sultan Qaboos University (Other)
Responsible Party: Principal Investigator, Mohammed Al Alawi MD PhD MRCPsych ARABpsych OMSBpsych, Assistant Professor, Sultan Qaboos University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 135
Record Dates: First submitted 2024-10-12; First posted 2024-10-16 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-10

CONDITIONS: Major Depressive Disorder
Keywords: Transcranial Magnetic Stimulation,; Antidepressants; iTMS; rTMS
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Transcranial Magnetic Stimulation; Antidepressive Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Transcranial magnetic stimulation (Experimental): Participants will receive repetitive Transcranial Magnetic Stimulation (rTMS) sessions, targeting the dorsolateral prefrontal cortex, at a frequency of 10 Hz. Each session will last approximately 30 minutes, with 5 sessions per week for 4 to 6 weeks. TMS will be administered by certified professionals, and patients will be monitored for any adverse events during each session. Follow-up evaluations will occur at regular intervals over the 3-year study period.
  Interventions: Device: Transcranial magnetic stimulation
- Treatment as usual (Active Comparator): Participants in this group will continue receiving standard care, which includes pharmacological management and psychotherapy based on clinical standards for MDD. Common medications may include selective serotonin reuptake inhibitors (SSRIs) or tricyclic antidepressants, with dose adjustments made based on clinical response. Psychotherapy will involve cognitive-behavioral therapy or supportive therapy sessions as determined by the attending psychiatrist.
  Interventions: Drug: Antidepressant

INTERVENTIONS:
Device: Transcranial magnetic stimulation — Transcranial Magnetic Stimulation (rTMS) sessions, targeting the dorsolateral prefrontal cortex, at a frequency of 10 Hz. Each session will last approximately 30 minutes, with 5 sessions per week for 4 to 6 weeks.
  Arms: Transcranial magnetic stimulation
Drug: Antidepressant — Selective serotonin reuptake inhibitors (SSRIs) or tricyclic antidepressants, SNRIs
  Arms: Treatment as usual

SUMMARY:
This clinical trial aims to assess the effectiveness of Transcranial Magnetic Stimulation (TMS) compared to Treatment as Usual (TAU) in adult patients experiencing their first or second episode of unipolar major depressive disorder (MDD). The primary end point is to determine whether TMS leads to higher rate of remission, response and greater reductions in depression severity, and improved functional outcomes compared to standard pharmacological and psychotherapeutic interventions. The trial will also explore the impact of TMS on quality of life and anxiety symptoms. Participants will be randomly assigned to either the TMS or TAU group, and outcomes will be assessed at multiple time points over a 3-year period. The trial will be conducted at Sultan Qaboos University Hospital's Department of Behavioural Medicine in Muscat, Oman, and is expected to contribute important evidence on the role of non-invasive brain stimulation in treating early-stage depression.

DETAILED DESCRIPTION:
1.1. Background and Rationale First-episode depression (FED) comprises 50% of major depressive disorder (MDD) cases in the U.S. and contributes 80% of global disability due to mental and substance use disorders. Depression significantly impairs social and occupational functioning, ranking third among the leading causes of global disease burden for individuals aged 10-65. Untreated, FED may progress to chronic depression, addiction, and increased healthcare costs. Given the limitations of current antidepressant treatments, there is a growing need for alternative interventions, such as transcranial magnetic stimulation (TMS). TMS is a non-invasive, well-accepted therapy with emerging evidence of efficacy for depression, but its use in first-episode depression requires further research. This trial aims to compare the effectiveness of TMS versus Treatment as Usual (TAU) for adult FED patients.

1.2. Study Scope This open-label study will follow FED patients (≥18 years) with moderate or severe MDD in an outpatient setting. Exclusion criteria include substance abuse, psychotic or catatonic features, suicidal risk, or previous ineffective TMS treatment. Pregnant or breastfeeding women can participate with neurologist approval. Primary outcomes will measure depression severity and functional impairment, assessed at baseline and at four key follow-up points.

2. Methodology A randomized controlled trial (RCT) will assess the comparative effectiveness of TMS and TAU. Participants will be randomly assigned to receive either TMS or TAU, with depression severity measured by standardized scales such as the Hamilton Depression Rating Scale (HAMD-24) and the World Health Organization Disability Assessment Schedule (WHO-DAS 2.0). Baseline data and follow-up assessments will evaluate the impact of treatment on depressive symptoms, quality of life, and functional outcomes.

2.1. Study Design The study will recruit adult patients experiencing their first episode of MDD. Inclusion and exclusion criteria will ensure a homogenous sample. Participants will provide written informed consent and undergo baseline assessments before randomization into either the TMS or TAU group. TMS will be administered by trained operators using a standardized protocol. Follow-up will occur over six months, with assessments of depressive symptoms, functional outcomes, and quality of life at regular intervals.

2.2. Interventions Participants in the TMS group will receive 10 Hz stimulation at 120% motor threshold for ≤30 minutes per session. The TAU group will follow standard pharmacological and psychotherapeutic management. Safety measures include constant monitoring during TMS sessions, with anxiety management protocols in place.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18 years old till 64 years) diagnosed with a first or second episode of unipolar major depressive disorder (MDD).
* Moderate to severe depressive symptoms based on clinical assessment and validated scales (e.g., Hamilton Depression Rating Scale (HDRS)).
* Willingness to participate and provide written informed consent.
* Outpatient setting (not currently hospitalized for psychiatric reasons).

Exclusion Criteria:

* Current episode is not the first or second episode of MDD.
* Substance dependence or abuse within the last 6 months.
* Diagnosed with psychotic depression, bipolar disorder, or catatonic features.
* Severe depression requiring electroconvulsive therapy (ECT).
* High suicidal risk as determined by clinical assessment.
* History of unsatisfactory responses to prior TMS treatments.
* Diagnosis of Epilepsy and Epilepsy high risk group
* Pregnant or breastfeeding women, unless cleared by a neurologist for TMS treatment.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2028-12-30 (Estimated); Study Completion 2029-06-01 (Estimated)

PRIMARY OUTCOMES:
Remission and Response rates between the two arms | 6 weeks
  Hamilton Depression Rating Scale (HDRS) The Hamilton Depression Rating Scale (HDRS) is a clinician-administered questionnaire commonly used to assess the severity of depression. It consists of 17 to 21 items, depending on the version used. Each item is scored on a scale from 0 to 2 or 0 to 4, with higher scores indicating more severe depression.
  Minimum Score: 0
  Maximum Score: 52 (for the 17-item version) or 64 (for the 21-item version)
  Interpretation: Higher scores reflect greater severity of depressive symptoms, with cut-offs typically used to classify depression as mild, moderate, severe, or very severe.
Remission and Response rates between the two arms | 6 weeks
  Patient Health Questionnaire-9 (PHQ-9) The PHQ-9 is a self-administered scale used to assess the severity of depression. It consists of 9 items that correspond to the diagnostic criteria for major depressive disorder (MDD) in the DSM-5. Each item is scored from 0 ("Not at all") to 3 ("Nearly every day").
  Minimum Score: 0
  Maximum Score: 27
  Interpretation: Higher scores indicate more severe depressive symptoms. Scores are often interpreted as follows:
  0-4: None to minimal depression
  5-9: Mild depression
  10-14: Moderate depression
  15-19: Moderately severe depression
  20-27: Severe depression
Remission and Response rates between the two arms | 6 weeks
  Quick Inventory of Depressive Symptomatology - Self-Report (QIDS-SR) The QIDS-SR is a brief, 16-item self-report questionnaire designed to assess the severity of depressive symptoms over the past week. Each item is scored on a scale from 0 to 3.
  Minimum Score: 0
  Maximum Score: 27
  Interpretation: Higher scores indicate more severe depression. Scores are typically classified as:
  0-5: Normal (no depression)
  6-10: Mild depression
  11-15: Moderate depression
  16-20: Severe depression
  21-27: Very severe depression

SECONDARY OUTCOMES:
Change in the Means Scores between the two arms at the end of the study of the GAD-7 andWHO-DAS 2.0) | 6 weeks
  ---
  WHO Disability Assessment Schedule (WHO-DAS 2.0) - 12-item Version The WHO-DAS 2.0 is a tool developed by the World Health Organization to measure health and disability across six domains: cognition, mobility, self-care, getting along with others, life activities, and participation in society. The 12-item version is a shortened version of the 36-item scale, designed for easier use while still covering the key aspects of disability. Each item is scored on a scale from 1 ("None") to 5 ("Extreme or cannot do").
  Minimum Score: 12
  Maximum Score: 60
  Interpretation: Higher scores indicate greater levels of disability. The total score can also be converted to a percentage (0-100), with higher percentages reflecting greater disability. This version provides a quick overview of an individual's level of functioning across multiple domains.
  ---
Change in the Means Scores between the two arms at the end of the study of the GAD-7 andWHO-DAS 2.0) | 6 weeks
  Generalized Anxiety Disorder-7 (GAD-7) The GAD-7 is a brief, self-report questionnaire used to assess the severity of generalized anxiety disorder (GAD). It consists of 7 items that ask respondents to rate how often they have been bothered by various anxiety symptoms over the past two weeks. Each item is scored from 0 ("Not at all") to 3 ("Nearly every day").
  Minimum Score: 0
  Maximum Score: 21
  Interpretation: Higher scores indicate more severe anxiety. Scores are typically classified as follows:
  0-4: Minimal anxiety
  5-9: Mild anxiety
  10-14: Moderate anxiety
  15-21: Severe anxiety